CLINICAL TRIAL: NCT01668719
Title: A Randomized Phase I/II Study of Optimal Induction Therapy of Bortezomib, Dexamethasone and Lenalidomide With or Without Elotuzumab (NSC-764479) for Newly Diagnosed High Risk Multiple Myeloma (HRMM)
Brief Title: S1211 Bortezomib, Dexamethasone, and Lenalidomide With or Without Elotuzumab in Treating Patients With Newly Diagnosed High-Risk Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1211; NCI-2012-01998 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PS1211_A12PAMDREVW01; CDR0000738512; S1211 (Other: SWOG); S1211 (Other: CTEP); U10CA180888 (NIH); U10CA032102 (NIH)
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Results first posted 2021-10-27 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: DS Stage I Plasma Cell Myeloma; DS Stage II Plasma Cell Myeloma; DS Stage III Plasma Cell Myeloma
MeSH Terms: interventions — Bortezomib; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; elotuzumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (bortezomib, lenalidomide, dexamethasone) (Active Comparator): INDUCTION: Patients receive bortezomib SC or IV on days 1, 4, 8, and 11; lenalidomide PO QD on days 1-14; and dexamethasone PO or IV on days 1, 2, 4, 5, 8, 9, 11, and 12. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity (patients who received a course of chemotherapy prior to registration will begin protocol treatment with course 2 and receive a total of 7 courses of protocol therapy).
  MAINTENANCE: Patients receive bortezomib SC or IV on days 1, 8, and 15; lenalidomide PO QD on days 1-21; and dexamethasone PO on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide
- Arm II (bortezomib, lenalidomide, dexamethasone, elotuzumab) (Experimental): INDUCTION: Patients receive bortezomib, lenalidomide, and dexamethasone as in Arm I. Patients also receive elotuzumab IV on days 1, 8, and 15 of courses 1 and 2 and on days 1 and 11 of courses 3-8. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive bortezomib, lenalidomide, and dexamethasone as in Arm I. Patients also receive elotuzumab IV on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Biological: Elotuzumab; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide

INTERVENTIONS:
Drug: Bortezomib — Given SC or IV
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Biological: Elotuzumab — Given IV
  Other Names: BMS-901608; HuLuc63; PDL-063; PDL063
  Arms: Arm II (bortezomib, lenalidomide, dexamethasone, elotuzumab)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid

SUMMARY:
This partially randomized phase I/II trial studies the side effects and best dose of elotuzumab and to see how well it works when given together with lenalidomide, bortezomib, and dexamethasone in treating patients with newly diagnosed multiple myeloma that is likely to recur (come back), or spread (high-risk). Lenalidomide and bortezomib may stop the growth of multiple myeloma by blocking blood flow to the tumor. Also, bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as lenalidomide and dexamethasone, also work in different ways to kill cancer cells, by stopping them from dividing, or by stopping them from spreading. Giving elotuzumab together with lenalidomide, bortezomib, and dexamethasone may be a better way to block cancer growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the appropriate Phase II dose of elotuzumab to use in combination with lenalidomide, bortezomib, and dexamethasone for patients with multiple myeloma. (Phase I) II. To assess whether incorporation of the novel agent elotuzumab into the treatment algorithm of high-risk multiple myeloma (HRMM) will improve progression-free survival (PFS). (Phase II) III. To estimate the frequency and severity of toxicities of this treatment strategy in this patient population. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of elotuzumab, followed by a phase II, randomized study.

PHASE I:

INDUCTION: Patients receive bortezomib subcutaneously (SC) or intravenously (IV) on days 1, 4, 8, and 11; lenalidomide orally (PO) once daily (QD) on days 1-14; and dexamethasone PO or IV on days 1, 2, 4, 5, 8, 9, 11, and 12 (and on day 15 of courses 1 and 2 only). Patients also receive elotuzumab IV on days 1, 8, and 15 of courses 1 and 2 and on days 1 and 11 of courses 3-8. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive bortezomib SC or IV on days 1, 8, and 15; lenalidomide PO QD on days 1-21; dexamethasone PO on days 1, 8, and 15; and elotuzumab IV on days 1 and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 treatment arms.

ARM I:

INDUCTION: Patients receive bortezomib SC or IV on days 1, 4, 8, and 11; lenalidomide PO QD on days 1-14; and dexamethasone PO or IV on days 1, 2, 4, 5, 8, 9, 11, and 12. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity (patients who received a course of chemotherapy prior to registration will begin protocol treatment with course 2 and receive a total of 7 courses of protocol therapy).

MAINTENANCE: Patients receive bortezomib SC or IV on days 1, 8, and 15; lenalidomide PO QD on days 1-21; and dexamethasone PO on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II:

INDUCTION: Patients receive bortezomib, lenalidomide, and dexamethasone as in Arm I. Patients also receive elotuzumab IV on days 1, 8, and 15 of courses 1 and 2 and on days 1 and 11 of courses 3-8. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive bortezomib, lenalidomide, and dexamethasone as in Arm I. Patients also receive elotuzumab IV on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed active multiple myeloma (MM)
* For the Phase II portion only, patients must have high-risk MM based on one or more of the following criteria at the time of initial diagnosis (prior to any chemotherapy):

  * Poor-risk genomic signature according to the University of Arkansas 70-gene model (available clinically as myeloma prognostic risk score [MyPRS] score, Signal Genetics, Inc) AND/OR
  * Translocation (14;16), and/or translocation (14;20), and/or deletion (17p) by fluorescence in-situ hybridization (FISH) or cytogenetics AND/OR
  * Primary plasma cell leukemia (defined by either >= 2,000 plasma cells/mL of peripheral blood, or 20% on a manual differential count) AND/OR
  * Serum lactate dehydrogenase (LDH) >= 2 x institutional upper limit of normal (IULN) AND/OR
  * 1q21 amplification by FISH analysis AND/OR
  * High risk by the SKY92 signature
* Patients with non-secretory MM or known amyloidosis are not eligible
* Patients must have measurable disease within 28 days prior to registration (or prior to initiation of first induction course for patients with prior therapy)
* Patients on the Phase I portion may not have received ANY prior chemotherapy; patients on the Phase II portion may have received one prior cycle of any non-investigational chemotherapy; prior chemotherapy must have been completed within 56 days prior to registration and all toxicities must have resolved to =< grade 1; patients on either portion may have received prior treatment with dexamethasone, providing total number of days of treatment was =< 14 days and total treatment dose was =< 360 mg
* Patients may have received prior radiotherapy for symptomatic localized bone lesions or impending spinal cord compression only; radiotherapy must be completed at least 14 days prior to registration and all toxicities must have resolved to =< grade 1
* Absolute neutrophil count (ANC) >= 1,000 cells/mm^3 without growth factor support
* Platelet count >= 70,000 cells/mm^3 for patients who have bone marrow plasmacytosis < 50%; or >= 50,000 cells/mm^3 for patients who have bone marrow plasmacytosis of >= 50%
* Total bilirubin =< 1.5 x institutional upper limit of normal (IULN)
* Serum glutamic oxaloacetic transaminase (SGOT)/aspartate aminotransferase (AST) and serum glutamate pyruvate transaminase (SGPT)/alanine aminotransferase (ALT) =< 2.5 x IULN
* Creatinine clearance (CrCL) >= 30 mL/min, measured by a 24-hour urine collection or estimated by the Cockcroft and Gault formula within 14 days prior to registration
* Patients must not have active involvement of the central nervous system (CNS) with MM (by clinical evaluation); patients with documentation of, or clinical signs or symptoms consistent with, CNS involvement of MM must have a lumbar puncture that is negative for CNS involvement of MM; the lumbar puncture must be completed within 14 days prior to registration; patients with no previous history of documented CNS involvement and with no clinical signs or symptoms consistent with CNS involvement are not required to have completed a lumbar puncture prior to registration; note that monitoring of CNS involvement and treatment with intrathecal therapy is recommended during protocol treatment
* Patients who are known to be human immunodeficiency virus positive (HIV+) are eligible providing they meet all of the following additional criteria within 28 days prior to registration:

  * Cluster of differentiation (CD)4 cells >= 500/mm^3
  * Viral load of < 50 copies HIV messenger ribonucleic acid (mRNA)/mm^3 if on combination antiretroviral therapy (cART) or < 25,000 copies HIV mRNA if not on cART
  * No zidovudine or stavudine as part of cART
  * Patients who are HIV+ and do not meet all of these criteria are not eligible for this study
* Patients must have baseline skeletal survey (whole body x-ray) to document lytic lesions, osteopenia or compression fracture
* Patients must have Zubrod performance status =< 2
* Patients with known hepatitis B or hepatitis C infection may be eligible providing they have viral load < 800,000 IU/L within 28 days prior to registration
* Patients must not have POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Patients must not have clinically significant illness including uncontrolled, active infection requiring intravenous antibiotics, New York Heart Association (NYHA) class III or class IV heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled >= grade 3 cardiac arrhythmias, uncontrolled hypertension, or uncontrolled diabetes mellitus; patients must have undergone an electrocardiogram (EKG) within 28 days prior to registration
* Uncontrolled diabetes: a glycated hemoglobin (Hg A1C) > 7% within 14 days prior to registration; the same criterion will be used in patients with confirmed diagnosis of diabetes mellitus who have been on a stable dietary or therapeutic regimen for this condition in the last three months
* Uncontrolled blood pressure and hypertension: systolic blood pressure (SBP) > 140 mm Hg or diastolic blood pressure (DBP) > 90 mm Hg within 14 days prior to registration; patients are permitted to be receiving multiple anti-hypertensive medications (unless otherwise indicated in the study); all blood pressure measurements within the 14 days prior to registration and on day 1 of cycle 1 must be SBP =< 140 and DBP =< 90; an exception can be made by a healthcare provider for a patient with a single blood pressure elevation who upon rechecking has a normal blood pressure
* Patients must have history and physical examination within 28 days prior to registration
* Patients must not have any psychiatric illness that could potentially interfere with the completion of treatment according to this protocol
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to registration; (Note: that pregnancy testing is also required within 24 hours prior to treatment on cycle 1, day 1); furthermore, they must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control: one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before starting lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP, even if they have had a successful vasectomy; a FCBP is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years
* Patients must be offered participation in banking of specimens for future research; with the patient's consent, specimens (serum and bone marrow biopsy core) must be submitted to the repository; patient consent must be obtained before specimens are submitted
* Patients must be registered to the mandatory Revlimid Risk Evaluation and Mitigation Strategy (REMS)™ program and must be willing and able to comply with the requirements of the Revlimid REMS™ program
* Patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2012-11; Primary Completion 2020-02-05 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Saad Usmani, Principal Investigator — SWOG Cancer Research Network
Locations (417):
- United States (417):
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Medical Oncology and Hematology Group PC-Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Charlotte Hungerford Hospital Center for Cancer Care, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Hines Veterans Administration Hospital, Hines, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Newman Regional Health, Emporia, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Olathe Medical Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Hematology/Oncology Clinic LLP, Baton Rouge, Louisiana
  - West Jefferson Medical Center, Marrero, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Community Hospital, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Providence Hospital-Southfield Cancer Center, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center-Carrie J Babb Cancer Center, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - CoxHealth Cancer Center, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-North, Kansas City, Missouri
  - The University of Kansas Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Faith Regional Medical Offices West, Norfolk, Nebraska
  - Great Plains Regional Medical Center, North Platte, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Oncology Hematology West, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Urology Cancer Center PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Regional West Medical Center, Scottsbluff, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - 21st Century Oncology - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology - Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Nevada Cancer Specialists-Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - 21st Century Oncology - Vegas Tenaya, Las Vegas, Nevada
  - Orange Regional Medical Center, Middletown, New York
  - University of Rochester, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Carolinas HealthCare System NorthEast, Concord, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Carolinas HealthCare System Union, Monroe, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hosiptal, Pinehurst, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Cleveland Clinic Cancer Center Beachwood, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geaugra Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OneHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Ireland Cancer Center Landerbrook Health Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Ireland Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH-Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Geisinger Medical Oncology-Pottsville, Pottsville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - M D Anderson Cancer Center, Houston, Texas
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Memorial Hospital Of Martinsville, Martinsville, Virginia
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic-Marinette, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Lakeview Medical Center-Marshfield Clinic, Rice Lake, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Derived] Banerjee R, Sexton R, Cowan AJ, Rosenberg AS, Ailawadhi S, Rajkumar SV, Kumar S, Dispenzieri A, Lonial S, Durie BGM, Richardson PG, Usmani SZ, Hoering A, Orlowski RZ. Dexamethasone dose intensity does not impact outcomes in newly diagnosed multiple myeloma: a secondary SWOG analysis. Blood. 2025 Jan 2;145(1):75-84. doi: 10.1182/blood.2024025939. PMID 39321347
- [Derived] Usmani SZ, Hoering A, Ailawadhi S, Sexton R, Lipe B, Hita SF, Valent J, Rosenzweig M, Zonder JA, Dhodapkar M, Callander N, Zimmerman T, Voorhees PM, Durie B, Rajkumar SV, Richardson PG, Orlowski RZ; SWOG1211 Trial Investigators. Bortezomib, lenalidomide, and dexamethasone with or without elotuzumab in patients with untreated, high-risk multiple myeloma (SWOG-1211): primary analysis of a randomised, phase 2 trial. Lancet Haematol. 2021 Jan;8(1):e45-e54. doi: 10.1016/S2352-3026(20)30354-9. Epub 2020 Dec 22. PMID 33357482

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 8 participants were enrolled to the Phase 1 Level 1 dose arm. 2 were ineligible, so 6 participants were assessed for DLT.
  In Phase II, 68 participants were enrolled on RVD and 66 to RVD/Elo arm. of these, 16 and 18 respectively were ineligible. Thus, 52 participants on RVD and 48 participants on RVD/Elo arm were eligible and evaluable for analyses.
Groups:
- Phase I Dose Level 1 (Elotuzumab, 10mg, and Bortezomib, Lenalidomide and Dexamethasone): INDUCTION: Participants receive bortezomib subcutaneously (SC) or intravenously (IV) on days 1, 4, 8, and 11; lenalidomide orally (PO) once daily (QD) on days 1-14; and dexamethasone PO or IV on days 1, 2, 4, 5, 8, 9, 11, and 12 (and on day 15 of courses 1 and 2 only). Participants also receive elotuzumab IV on days 1, 8, and 15 of courses 1 and 2 and on days 1 and 11 of courses 3-8. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Participants receive bortezomib SC or IV on days 1, 8, and 15; lenalidomide PO QD on days 1-21; dexamethasone PO on days 1, 8, and 15; and elotuzumab IV on days 1 and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm I (Bortezomib, Lenalidomide, Dexamethasone): INDUCTION: Participants receive bortezomib SC or IV on days 1, 4, 8, and 11; lenalidomide PO QD on days 1-14; and dexamethasone PO or IV on days 1, 2, 4, 5, 8, 9, 11, and 12. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity (participants who received a course of chemotherapy prior to registration will begin protocol treatment with course 2 and receive a total of 7 courses of protocol therapy).
  MAINTENANCE: Participants receive bortezomib SC or IV on days 1, 8, and 15; lenalidomide PO QD on days 1-21; and dexamethasone PO on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Bortezomib: Given SC or IV
  Dexamethasone: Given PO or IV
  Laboratory Biomarker Analysis: Correlative studies
  Lenalidomide: Given PO
- Arm II (Bortezomib, Lenalidomide, Dexamethasone, Elotuzumab): INDUCTION: Participants receive bortezomib, lenalidomide, and dexamethasone as in Arm I. Participants also receive elotuzumab IV on days 1, 8, and 15 of courses 1 and 2 and on days 1 and 11 of courses 3-8. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Participants receive bortezomib, lenalidomide, and dexamethasone as in Arm I. Participants also receive elotuzumab IV on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Bortezomib: Given SC or IV
  Dexamethasone: Given PO or IV
  Elotuzumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Lenalidomide: Given PO
Period: Phase I
Arm/Group | Phase I Dose Level 1 (Elotuzumab, 10mg, and Bortezomib, Lenalidomide and Dexamethasone) | Arm I (Bortezomib, Lenalidomide, Dexamethasone) | Arm II (Bortezomib, Lenalidomide, Dexamethasone, Elotuzumab)
Started | 6 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 6 | 0 | 0
Not completed — On treatment | 1 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Progression/relapse | 1 | 0 | 0
Not completed — not protocol specified | 2 | 0 | 0
Period: Phase II
Arm/Group | Phase I Dose Level 1 (Elotuzumab, 10mg, and Bortezomib, Lenalidomide and Dexamethasone) | Arm I (Bortezomib, Lenalidomide, Dexamethasone) | Arm II (Bortezomib, Lenalidomide, Dexamethasone, Elotuzumab)
Started | 0 | 52 | 48
Completed | 0 | 0 | 0
Not Completed | 0 | 52 | 48
Not completed — On treatment | 0 | 4 | 3
Not completed — Adverse Event | 0 | 18 | 18
Not completed — Refusal unrelated to adverse event | 0 | 4 | 1
Not completed — Progression/relapse | 0 | 13 | 17
Not completed — Death | 0 | 0 | 2
Not completed — not protocol specified | 0 | 13 | 7

BASELINE CHARACTERISTICS:
Population: All eligible participants
Groups:
- Arm II (Bortezomib, Lenalidomide, Dexamethasone, Elotuzumab): INDUCTION: Participants receive bortezomib, lenalidomide, and dexamethasone as in Arm I. Participants also receive elotuzumab IV on days 1, 8, and 15 of courses 1 and 2 and on days 1 and 11 of courses 3-8. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE:Participants receive bortezomib, lenalidomide, and dexamethasone as in Arm I. Participants also receive elotuzumab IV on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Bortezomib: Given SC or IV
  Dexamethasone: Given PO or IV
  Elotuzumab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Lenalidomide: Given PO
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Level 1 (Elotuzumab, 10mg, and Bortezomib, Lenalidomide and Dexamethasone) | Arm I (Bortezomib, Lenalidomide, Dexamethasone) | Arm II (Bortezomib, Lenalidomide, Dexamethasone, Elotuzumab) | Total
Number analyzed (Participants) | 6 | 52 | 48 | 106
Age, Continuous [Median (Full Range); unit: years] | 67.6 [56.1 to 79.3] | 65.6 [36.1 to 84.5] | 62.3 [40.0 to 78.6] | 64.2 [36.1 to 84.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 21 | 19 | 43
  Male | 3 | 31 | 29 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 3
  Not Hispanic or Latino | 5 | 48 | 45 | 98
  Unknown or Not Reported | 0 | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 8 | 6 | 15
  White | 3 | 44 | 41 | 88
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 1 | 3
PCL and/or high LDH [Count of Participants; unit: Participants] — PCL- plasma cell leukemia LDH- lactate dehydrogenase
  Participants
    Yes | 1 | 9 | 6 | 16
    No | 5 | 43 | 42 | 90

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of Elotuzumab in Combination With Bortezomib, Lenalidomide and Dexamethasone
Description: Assess safety of elotuzumab in combination with bortezomib, lenalidomide and dexamethasone and select the optimal dose of elotuzumab for the Phase II portion from 10mg/kg on each cycle, to 5mg/kg on each cycle MTD reflects the highest dose that had a dose-limiting toxicity (DLT) rate of ≤ 1/6 participants. DLTs were defined as treatment regimen related: grade ≥ 3 non-hematologic toxicity; grade 3 nausea or diarrhea despite anti-emetic and anti-diarrheal therapy; grade 3 hyperglycemia if symptomatic or glucose level > 300mg/ml despite insulin and/or oral diabetic therapy; grade 4 neutropenia ≥ 7 days or grade 3/4 neutropenia with fever (≥ 38.5 oC); grade 4 thrombocytopenia ≥ 7 days or associated with hemorrhage; delay of treatment with any agent by > 2 weeks due to drug related toxicity.
  DLT were graded using the NCI CTCAE version 4.0
  Note:
  i) the second, lower dose level was not tested as the first dose level was deemed safe ii) 6 participants were evaluable at phase I analysis
Time Frame: time from first participants randomized until at least 6 patients were evaluable for DLTs. DLTs were assessed only during Cycle 1 (21 days)
Population: At the time of the phase I analysis, six participants were evaluable for DLTs (i.e. were eligible and received at least one dose of study drug).
Measure: Number; unit: mg/kg (Phase II dosing for elotuzumab)
Arm/Group | Phase I Dose Level 1 (Elotuzumab, 10mg, and Bortezomib, Lenalidomide and Dexamethasone)
Number analyzed (Participants) | 6
mg/kg (Phase II dosing for elotuzumab) | 10

2. Primary Outcome: Progression-free Survival
Description: From date of registration to date of first documentation of progression or death due to any cause.
  Per the International Uniform Response Criteria for Multiple Myeloma, progression is defined as >=1 of Serum M protein increase >= 25% from lowest response level, with an absolute increase of >= 0.5g/dL; Urine M protein increase >= 25% from lowest response level, with an absolute increase of >= 200 mg/24 hrs; If participant had serum M protein <1 g/dL, urine M protein <200 mg/24 hrs, and an involved serum free light chain level >= 10mg/dL at baseline: >= 25% increase in the difference between involved and uninvolved serum free light chain level with an absolute increase of >= 10 mg/dL; Bone marrow plasma cell % increase =25% from baseline with the absolute plasma cell % >=10%; New bone lesions or soft tissue plasmocytomas, or definite increase in size of existing bone lesions or soft tissue plasmocytomas; Development of hypercalcemia that can be attributed solely to multiple myeloma
Time Frame: Up to 6 years post registration
Population: Eligible and analyzable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Bortezomib, Lenalidomide, Dexamethasone) | Arm II (Bortezomib, Lenalidomide, Dexamethasone, Elotuzumab)
Number analyzed (Participants) | 52 | 48
months | 33.6 [19.6 to NA] — not reached | 31.5 [18.6 to 54.0]

3. Secondary Outcome: Number of Participants With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Adverse Events (AEs) are reported by CTCAE Version 4.0. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Duration of treatment and follow up until death or 6 years post registration, whichever occurs first.
Population: Participants who received at least one dose of protocol treatment.
Measure: Number; unit: Participants
Groups:
- Arm I (Bortezomib, Lenalidomide, Dexamethasone): INDUCTION: Participants receive bortezomib SC or IV on days 1, 4, 8, and 11; lenalidomide PO QD on days 1-14; and dexamethasone PO or IV on days 1, 2, 4, 5, 8, 9, 11, and 12. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity (participants who received a course of chemotherapy prior to registration will begin protocol treatment with course 2 and receive a total of 7 courses of protocol therapy).
  MAINTENANCE: Participants receive bortezomib SC or IV on days 1, 8, and 15; lenalidomide PO QD on days 1-21; and dexamethasone PO on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Bortezomib: Given SC or IV
  Dexamethasone: Given PO or IV
  Lenalidomide: Given PO
- Arm II (Bortezomib, Lenalidomide, Dexamethasone, Elotuzumab): INDUCTION: Participants receive bortezomib, lenalidomide, and dexamethasone as in Arm I. Participants also receive elotuzumab IV on days 1, 8, and 15 of courses 1 and 2 and on days 1 and 11 of courses 3-8. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Participants receive bortezomib, lenalidomide, and dexamethasone as in Arm I. Participants also receive elotuzumab IV on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Bortezomib: Given SC or IV
  Dexamethasone: Given PO or IV
  Elotuzumab: Given IV
  Lenalidomide: Given PO
Arm/Group | Arm I (Bortezomib, Lenalidomide, Dexamethasone) | Arm II (Bortezomib, Lenalidomide, Dexamethasone, Elotuzumab)
Number analyzed (Participants) | 52 | 48
Participants
  Abdominal pain | 1 | 0
  Acute kidney injury | 1 | 0
  Agitation | 0 | 1
  Alanine aminotransferase increased | 0 | 2
  Alkaline phosphatase increased | 0 | 1
  Allergic reaction | 0 | 1
  Anemia | 8 | 6
  Aspartate aminotransferase increased | 0 | 2
  Atrial fibrillation | 3 | 0
  Back pain | 0 | 1
  Blood bilirubin increased | 0 | 1
  Bone pain | 0 | 2
  Cataract | 0 | 1
  Creatinine increased | 0 | 1
  Diarrhea | 5 | 1
  Dizziness | 1 | 0
  Dry skin | 1 | 0
  Dyspnea | 0 | 2
  Edema limbs | 2 | 0
  Encephalopathy | 1 | 0
  Eye disorders - Other, specify | 0 | 1
  Fall | 1 | 0
  Fatigue | 6 | 5
  Febrile neutropenia | 2 | 1
  Fracture | 0 | 1
  Gait disturbance | 1 | 0
  Gastrointestinal disorders - Other, specify | 0 | 1
  Generalized muscle weakness | 1 | 1
  Hyperglycemia | 2 | 4
  Hyperkalemia | 1 | 1
  Hypertension | 2 | 1
  Hypoalbuminemia | 0 | 1
  Hypokalemia | 0 | 4
  Hyponatremia | 3 | 1
  Hypophosphatemia | 1 | 0
  Hypotension | 2 | 4
  Hypoxia | 1 | 1
  INR increased | 0 | 1
  Infections and infestations - Other, specify | 3 | 4
  Infusion related reaction | 0 | 3
  Insomnia | 0 | 2
  Lung infection | 3 | 5
  Lymphocyte count decreased | 14 | 13
  Multi-organ failure | 0 | 1
  Muscle weakness lower limb | 2 | 0
  Muscle weakness trunk | 0 | 1
  Musculoskeletal and connective tiss disorder - Other | 1 | 0
  Nausea | 1 | 0
  Neck pain | 0 | 1
  Neuralgia | 0 | 1
  Neutrophil count decreased | 8 | 5
  Osteonecrosis of jaw | 1 | 0
  Pain | 0 | 1
  Pain in extremity | 1 | 0
  Peripheral motor neuropathy | 1 | 4
  Peripheral sensory neuropathy | 4 | 6
  Platelet count decreased | 10 | 10
  Pneumonitis | 0 | 1
  Portal vein thrombosis | 0 | 1
  Pulmonary edema | 1 | 0
  Rash acneiform | 1 | 0
  Rash maculo-papular | 2 | 3
  Resp, thoracic and mediastinal disorders - Other | 0 | 1
  Respiratory failure | 2 | 1
  Sepsis | 2 | 1
  Skin infection | 0 | 1
  Stroke | 0 | 1
  Supraventricular tachycardia | 0 | 1
  Syncope | 1 | 2
  Thromboembolic event | 4 | 1
  Tremor | 1 | 0
  Urinary tract infection | 2 | 0
  Urine output decreased | 0 | 1
  Vomiting | 1 | 0
  Weight loss | 0 | 1
  White blood cell decreased | 4 | 5

4. Secondary Outcome: Overall Survival
Description: From date of registration to date of death due to any cause
Time Frame: Up to 6 years post registration
Population: Eligible and evaluable participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Bortezomib, Lenalidomide, Dexamethasone) | Arm II (Bortezomib, Lenalidomide, Dexamethasone, Elotuzumab)
Number analyzed (Participants) | 52 | 48
months | NA [NA to NA] — median overall survival was not reached | 68 [61 to 68]

5. Secondary Outcome: Response (Partial Response [PR] or Better) Rate
Description: Percentage of participants with PR or better to treatment per the International Uniform Response Criteria for Multiple Myeloma stringent Complete Response- CR criteria + normal serum free light chain (FLC) ratio + absence of clonal cells in bone marrow (BM) by immunohistochemistry or immunofluorescence CR- Negative immunofixation (IFX) on serum & urine M proteins + <5% plasma cells in BM + disappearance of soft tissue plasmocytomas (STP) very good PR- PR criteria + serum & urine M proteins detectable by IFX but not on electrophoresis or >=90% reduction (RED) in serum M protein & urine M protein <100 g/24 hrs PR- >=50% RED in size of STP, if present at baseline & >=50% RED in plasma cells, if >=30% plasma cells in BM at baseline: & RED in serum M protein of >=50% & in urine M protein of >= 90% or to 200 mg/24hr OR if serum M protein <1 g/dL, urine M protein <200 mg/24 hrs, & involved serum FLC level >= 10 mg/dl at baseline: >= 50% RED in (involved-uninvolved) serum FLC levels
Time Frame: Up to 6 years post registration
Population: Eligible participants assessable for response at follow up. 1 participant on Arm II was not assessable for RR.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm I (Bortezomib, Lenalidomide, Dexamethasone) | Arm II (Bortezomib, Lenalidomide, Dexamethasone, Elotuzumab)
Number analyzed (Participants) | 52 | 47
Percentage of participants | 88 [76 to 95] | 83 [69 to 92]

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 6 years post registration, whichever occurs first.
Description: 6 participants in Phase I and 100 participants in Phase II were evaluable and assessed for AEs.
Groups:
- Phase I Dose Level 1 (Elotuzumab, 10mg, and Bortezomib, Lenali: INDUCTION: Participants receive bortezomib subcutaneously (SC) or intravenously (IV) on days 1, 4, 8, and 11; lenalidomide orally (PO) once daily (QD) on days 1-14; and dexamethasone PO or IV on days 1, 2, 4, 5, 8, 9, 11, and 12 (and on day 15 of courses 1 and 2 only). Participants also receive elotuzumab IV on days 1, 8, and 15 of courses 1 and 2 and on days 1 and 11 of courses 3-8. Treatment repeats every 21 days for 8 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Participants receive bortezomib SC or IV on days 1, 8, and 15; lenalidomide PO QD on days 1-21; dexamethasone PO on days 1, 8, and 15; and elotuzumab IV on days 1 and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Phase I Dose Level 1 (Elotuzumab, 10mg, and Bortezomib, Lenali | Arm I (Bortezomib, Lenalidomide, Dexamethasone) | Arm II (Bortezomib, Lenalidomide, Dexamethasone, Elotuzumab)
All-Cause Mortality (participants affected / at risk) | 2/6 | 19/52 | 16/48
Serious Adverse Events (participants affected / at risk) | 3/6 | 6/52 | 24/48
Other Adverse Events (participants affected / at risk) | 6/6 | 52/52 | 47/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level 1 (Elotuzumab, 10mg, and Bortezomib, Lenali (N=6) | Arm I (Bortezomib, Lenalidomide, Dexamethasone) (N=52) | Arm II (Bortezomib, Lenalidomide, Dexamethasone, Elotuzumab) (N=48)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1
Edema limbs (General disorders) | 0 | 0 | 2
Flu like symptoms (General disorders) | 0 | 0 | 1
Infusion related reaction (General disorders) | 0 | 0 | 2
Malaise (General disorders) | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 2
Infections and infestations-Other (Infections and infestations) | 1 | 1 | 5
Lung infection (Infections and infestations) | 0 | 0 | 7
Sepsis (Infections and infestations) | 0 | 1 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Creatinine increased (Investigations) | 0 | 0 | 1
INR increased (Investigations) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 4
Urine output decreased (Investigations) | 0 | 0 | 1
White blood cell decreased (Investigations) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Nervous system disorders-Other (Nervous system disorders) | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Stroke (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 3
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Erythroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1
Thromboembolic event (Vascular disorders) | 1 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level 1 (Elotuzumab, 10mg, and Bortezomib, Lenali (N=6) | Arm I (Bortezomib, Lenalidomide, Dexamethasone) (N=52) | Arm II (Bortezomib, Lenalidomide, Dexamethasone, Elotuzumab) (N=48)
Anemia (Blood and lymphatic system disorders) | 1 | 39 | 21
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 3 | 1
Cardiac disorders-Other (Cardiac disorders) | 1 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 2 | 0
Heart failure (Cardiac disorders) | 0 | 4 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 1
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 4 | 3
Sinus tachycardia (Cardiac disorders) | 0 | 2 | 4
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Ear and labyrinth disorders-Other (Ear and labyrinth disorders) | 1 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 3 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 3
Tinnitus (Ear and labyrinth disorders) | 2 | 3 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 1 | 0
Endocrine disorders-Other (Endocrine disorders) | 0 | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Blurred vision (Eye disorders) | 2 | 10 | 11
Cataract (Eye disorders) | 1 | 2 | 2
Conjunctivitis (Eye disorders) | 1 | 1 | 1
Dry eye (Eye disorders) | 0 | 2 | 2
Eye disorders-Other (Eye disorders) | 0 | 5 | 6
Flashing lights (Eye disorders) | 0 | 0 | 1
Floaters (Eye disorders) | 0 | 0 | 1
Optic nerve disorder (Eye disorders) | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 1 | 0
Scleral disorder (Eye disorders) | 0 | 1 | 0
Watering eyes (Eye disorders) | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 7 | 7
Bloating (Gastrointestinal disorders) | 1 | 2 | 3
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 37 | 24
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 5 | 29 | 24
Dry mouth (Gastrointestinal disorders) | 0 | 3 | 8
Dyspepsia (Gastrointestinal disorders) | 2 | 12 | 5
Dysphagia (Gastrointestinal disorders) | 0 | 4 | 5
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 2
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 | 7 | 6
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 0 | 4 | 3
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 2 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 6 | 6
Nausea (Gastrointestinal disorders) | 3 | 26 | 25
Oral pain (Gastrointestinal disorders) | 0 | 2 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 3 | 2
Toothache (Gastrointestinal disorders) | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 3 | 8 | 9
Chills (General disorders) | 3 | 9 | 8
Edema face (General disorders) | 0 | 4 | 3
Edema limbs (General disorders) | 6 | 33 | 29
Fatigue (General disorders) | 6 | 41 | 34
Fever (General disorders) | 3 | 11 | 13
Flu like symptoms (General disorders) | 4 | 0 | 3
Gait disturbance (General disorders) | 0 | 6 | 2
General disorders and admin site conditions - Other (General disorders) | 4 | 3 | 3
Infusion related reaction (General disorders) | 0 | 0 | 2
Infusion site extravasation (General disorders) | 0 | 0 | 1
Injection site reaction (General disorders) | 2 | 1 | 3
Irritability (General disorders) | 1 | 1 | 2
Localized edema (General disorders) | 0 | 4 | 1
Malaise (General disorders) | 0 | 3 | 2
Non-cardiac chest pain (General disorders) | 0 | 5 | 3
Pain (General disorders) | 3 | 14 | 14
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 1 | 2
Autoimmune disorder (Immune system disorders) | 1 | 0 | 0
Immune system disorders-Other (Immune system disorders) | 2 | 0 | 0
Bladder infection (Infections and infestations) | 1 | 0 | 0
Bronchial infection (Infections and infestations) | 2 | 2 | 1
Conjunctivitis infective (Infections and infestations) | 0 | 1 | 0
Endocarditis infective (Infections and infestations) | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 1
Gum infection (Infections and infestations) | 1 | 1 | 0
Infections and infestations-Other (Infections and infestations) | 3 | 11 | 5
Lung infection (Infections and infestations) | 0 | 7 | 4
Mucosal infection (Infections and infestations) | 1 | 1 | 2
Nail infection (Infections and infestations) | 0 | 0 | 1
Papulopustular rash (Infections and infestations) | 0 | 1 | 0
Peripheral nerve infection (Infections and infestations) | 0 | 1 | 0
Rhinitis infective (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 3 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 2
Skin infection (Infections and infestations) | 1 | 2 | 3
Soft tissue infection (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 5 | 8 | 8
Urinary tract infection (Infections and infestations) | 1 | 5 | 6
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 3 | 6
Burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 8 | 7
Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injury, poison and procedural complications - Other (Injury, poisoning and procedural complications) | 2 | 0 | 6
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 15 | 14
Alkaline phosphatase increased (Investigations) | 1 | 13 | 12
Aspartate aminotransferase increased (Investigations) | 1 | 9 | 10
Blood bilirubin increased (Investigations) | 1 | 6 | 1
Cholesterol high (Investigations) | 0 | 2 | 4
Creatinine increased (Investigations) | 1 | 14 | 9
Ejection fraction decreased (Investigations) | 0 | 1 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 1
Hemoglobin increased (Investigations) | 0 | 1 | 1
INR increased (Investigations) | 0 | 1 | 3
Investigations-Other (Investigations) | 1 | 1 | 0
Lymphocyte count decreased (Investigations) | 4 | 24 | 18
Lymphocyte count increased (Investigations) | 0 | 1 | 2
Neutrophil count decreased (Investigations) | 2 | 18 | 17
Platelet count decreased (Investigations) | 3 | 30 | 32
Weight gain (Investigations) | 1 | 8 | 11
Weight loss (Investigations) | 2 | 9 | 9
White blood cell decreased (Investigations) | 4 | 25 | 23
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 20 | 17
Dehydration (Metabolism and nutrition disorders) | 1 | 7 | 10
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 6 | 7
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 15 | 17
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 5 | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 6 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 15 | 20
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 21 | 21
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 6 | 7
Hypokalemia (Metabolism and nutrition disorders) | 2 | 18 | 18
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 6 | 5
Hyponatremia (Metabolism and nutrition disorders) | 2 | 14 | 14
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 6 | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 1 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 12 | 11
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 19 | 20
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 11 | 9
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 8 | 11
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 6 | 4
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 3 | 5 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 13 | 10
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 6
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 21 | 25
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Akathisia (Nervous system disorders) | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1 | 3
Cognitive disturbance (Nervous system disorders) | 0 | 1 | 0
Concentration impairment (Nervous system disorders) | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 3 | 22 | 19
Dysesthesia (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 13 | 10
Dysphasia (Nervous system disorders) | 0 | 0 | 2
Encephalopathy (Nervous system disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 2 | 16 | 14
Hypersomnia (Nervous system disorders) | 0 | 0 | 1
Ischemia cerebrovascular (Nervous system disorders) | 1 | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 2 | 6
Movements involuntary (Nervous system disorders) | 1 | 0 | 1
Nervous system disorders-Other (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 2
Paresthesia (Nervous system disorders) | 1 | 5 | 4
Peripheral motor neuropathy (Nervous system disorders) | 1 | 6 | 13
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 38 | 35
Presyncope (Nervous system disorders) | 0 | 2 | 2
Radiculitis (Nervous system disorders) | 1 | 4 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Sinus pain (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Spasticity (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 3 | 2
Tremor (Nervous system disorders) | 1 | 4 | 6
Agitation (Psychiatric disorders) | 0 | 1 | 4
Anxiety (Psychiatric disorders) | 2 | 8 | 10
Confusion (Psychiatric disorders) | 0 | 2 | 3
Depression (Psychiatric disorders) | 0 | 5 | 10
Insomnia (Psychiatric disorders) | 3 | 16 | 19
Personality change (Psychiatric disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 6 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 2
Hematuria (Renal and urinary disorders) | 0 | 1 | 3
Proteinuria (Renal and urinary disorders) | 0 | 4 | 4
Renal and urinary disorders-Other (Renal and urinary disorders) | 0 | 1 | 1
Renal calculi (Renal and urinary disorders) | 0 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 4 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 1 | 2
Urinary retention (Renal and urinary disorders) | 0 | 2 | 4
Urinary tract pain (Renal and urinary disorders) | 1 | 1 | 2
Urinary urgency (Renal and urinary disorders) | 0 | 1 | 1
Urine discoloration (Renal and urinary disorders) | 0 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 2 | 2
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 2
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 2 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 18 | 22
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 21 | 19
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 8 | 7
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 11
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Retinoic acid syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 7 | 8
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 5
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 3 | 7
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 6 | 6
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 3 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 18 | 12
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 6 | 5
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Surgical and medical procedures-Other (Surgical and medical procedures) | 1 | 1 | 2
Flushing (Vascular disorders) | 0 | 0 | 7
Hematoma (Vascular disorders) | 0 | 2 | 0
Hot flashes (Vascular disorders) | 0 | 2 | 6
Hypertension (Vascular disorders) | 1 | 21 | 17
Hypotension (Vascular disorders) | 1 | 13 | 14
Superficial thrombophlebitis (Vascular disorders) | 0 | 1 | 1
Thromboembolic event (Vascular disorders) | 2 | 6 | 6
Vascular disorders-Other (Vascular disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/19/NCT01668719/Prot_SAP_ICF_000.pdf